CLINICAL TRIAL: NCT07035548
Title: Design, Implementation, and Evaluation of Peer Learning in Teaching Technical Skills to Second-Year Nursing Students (
Brief Title: Design, Implementation, and Evaluation of Peer Learning in Teaching Technical Skills to Second-Year Nursing Students. (PL)
Acronym: (PL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marta Lizarbe (Other)
Responsible Party: Sponsor-Investigator, Marta Lizarbe, PhD, MsD, RNs, Clinica Universidad de Navarra, Universidad de Navarra
Organization: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2024.172
Record Dates: First submitted 2025-06-15; First posted 2025-06-25 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Urinary Catheterization; Simulation Training
Keywords: Peer-learning; procedural skills; urinary catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-learning (Experimental): Arm intervention group:
  Participants in the peer-learning intervention group will complete a structured educational program focused on acquiring urinary catheterization skills.
  The intervention includes:
  * (1) Self-Learning Preparation: Prior to the in-person session, participants will engage in general self-learning preparation (pre-briefing), completed independently outside the simulation center.
  * A two-hour in-person (2) Didactic Session will be dedicated to theoretical instruction and demonstration of urinary catheterization by a practical lecturer (ten minutes) and a peer-Guided Practice. Here, Students divided into pairs, will use a comprehensive guide for self-training and practice the procedural skills. This peer-supported practice allows for repeated attempts and immediate feedback. During the didactic session, participants are encouraged to practice as many times as necessary to achieve proficiency. Finally, and after peer-training, each participant's mastery of the skill w
  Interventions: Other: Educative: Peer-learning
- Traidional teaching (No Intervention): Arm control group:
  Participants in the control group will complete a structured educational program focused on acquiring urinary catheterization skills using traditional teaching methods, guided by a practical lecturer.
  The control group intervention includes: (1) Self-Learning Preparation: Prior to the in-person session, participants will engage in general self-learning preparation (pre-briefing), completed independently outside the simulation center. (2) Didactic Session: A two-hour in-person class dedicated to theoretical instruction and demonstration of urinary catheterization. A practical lecturer will demonstrate the procedure (20 minutes). There, students will individually practice the procedural skills, supported by the practical lecturer. This allows for repeated attempts and immediate feedback directly from the lecturer. (3) After completing their training, each participant's mastery of the skill will be formally evaluated by a qualified teacher.

INTERVENTIONS:
Other: Educative: Peer-learning — Peer learning, also known as peer-to-peer learning, is a collaborative educational strategy where students actively learn from one another. It involves interaction among peers to share knowledge, solve problems, and develop skills. This methodology can take various forms, from peer tutoring, where a more advanced student assists a less experienced one, to study groups where everyone contributes equally. The process fosters critical thinking, effective communication, and the co-construction of knowledge. By explaining concepts to others or discussing ideas, students solidify their own understanding and discover new perspectives. Moreover, it promotes individual and collective responsibility, as each participant plays an active role in their own learning and that of their peers. This approach not only improves academic performance but also develops crucial social and emotional skills, such as empathy, patience, and the ability to collaborate, preparing students for more cooperative work
  Arms: Peer-learning

SUMMARY:
The goal of this randomized controlled trial is to evaluate the effectiveness of a peer-learning educational intervention for teaching procedural skills to second-year nursing students. The study aims to answer the following key questions:

* Does the peer-learning intervention group gain equal or greater knowledge compared to those who learn by the traditional method?
* Do students in the peer-learning intervention group demonstrate higher self-efficacy for learning?
* Do students in the peer-learning intervention group demonstrate higher classroom engagement for learning?
* Do students in the peer-learning intervention group demonstrate higher general satisfaction with their learning experience?

Researchers will compare the peer-learning method with the traditional teaching methods to assess the acquisition of the procedural skill "urinary catheterization" in university nursing students.

Participants will:

* Attend a two-hour class to learn urinary catheterization.
* Work with a guide and a peer for self-training.
* Practice the procedural skills as many times as needed.
* Be evaluated by a teacher.

DETAILED DESCRIPTION:
Within the nursing curriculum, students dedicate significant effort to acquiring clinical procedural skills. Therefore, promoting student-centered educational activities with active learning methodologies fosters self-regulated learning and enhances commitment and participation in developing clinical competencies. Pedagogically grounded in social interaction and collaborative learning, as originally proposed by theorists like Piaget and Vygotsky, Peer-Learning has emerged as a valuable approach. Through this methodology, students learn by engaging in activities where they interact with peers, articulate their ideas and reflections, and practice giving and receiving feedback. As Joubert stated, "to teach is to learn twice."

Furthermore, it is crucial to assess each student's learning outcomes, their commitment to their own learning, and their satisfaction with the educational activity. This allows for reorientation or adaptation to specific educational contexts, ultimately leading to improved nursing training and a professional profile capable of meeting the current demands of healthcare.

General Objective

To design, implement, and evaluate the outcomes of implementing Peer-Learning for the nursing intervention of urinary catheterization among second-year nursing students.

ELIGIBILITY:
Inclusion Criteria:

* Second years nursing students

Exclusion Criteria:

* If participants have previously utilized peer learning as a method for acquiring or reinforcing knowledge and skills.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
General Knowledge | Immediatelly before and after the educative intervention.
  Each student's baseline knowledge will be assessed before participating in the Internship Experience (IE) Urinary catheterization. To do this, each student will complete an exam covering the content provided in the IE preparatory documentation (delivered via vitual educative platform, ADI) and from the lecture given to the entire class by a professor from the Practical Teaching Unit. The questionnaire, a multiple-choice test designed ad hoc by the researchers, will consist of 10 questions with four response options. Incorrect answers will not be penalized. The total possible score is 10 points. To prevent students from sharing exam content and to make memorization difficult, a bank of 30 questions has been created, from which different versions of the knowledge exam will be generated.
Self-Efficacy for learning clinical skills | Immediately after the intervention
  To measure the self-efficay with technical skills, the Learning Self-efficacy Scale for clinical skills (L-SES) was used. Developed by Kang et al. (2019), is a measurement instrument designed to understand the relationship between student self-efficacy and the practice of technical skills. This scale was developed under the framework of Bloom's Taxonomy and has been rigorously tested and validated in medical students. It demonstrated appropriate content validity indices (I-CVI = 0.88-1) and reliability (Cronbach's alpha of 0.931). Furthermore, results indicated that L-SES scores were not affected by gender (t = -0.049; 95% confidence interval [-,115; 0,109], p > 0.05). The L-SES comprises twelve items grouped into three distinct domains: cognitive, affective, and psychomotor. Responses are captured using a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree).
The engagement with learning | Immediately after the intervention
  The Learning Engagement Survey, developed by members of the Foundation for the Improvement of Postsecondary Education (U.S. Department of Education, 2003) is designed to measure students' self-perceived engagement with their learning during class. This survey consists of eight items grouped into two domains: Participation and Enjoyment. Responses are collected using a 5-point Likert scale (1 = strongly disagree; 2 = disagree; 3 = neither disagree nor agree; 4 = agree; 5 = strongly agree). The survey has demonstrated adequate validity and reliability, with an overall Cronbach's alpha of 0.881. The two subscales, Participation (five items) and Enjoyment (three items), yielded respective Cronbach's alpha values of 0.807 and 0.873 (Menenga et al., 2013).
Procedural skill | Immediately after the intervention
  To assess proficiency development in the procedural skill of urinary catheterization, students from both the intervention (peer-learning) and control (traditional teaching) groups were evaluated by an academic tutor. The tool developed was a 10-item rubric with a "yes/yes with changes/no" response format. The rubric underwent face and content validity with academic tutors. For consistency, the first six students were evaluated by two assessors, and any discrepancies were resolved by a third evaluator.

SECONDARY OUTCOMES:
General satisfaction | Just after the intervention
  To measure satisfaction, the General Satisfaction Survey with the Educational Activity, adapted from Hoseini et al. (2013) was used to collect information on student satisfaction with the training activity. This survey consists of 10 general satisfaction questions. Responses will be recorded using a 5-point Likert scale (1 = strongly disagree; 2 = disagree; 3 = neither disagree nor agree; 4 = agree; 5 = strongly agree).

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - University of Navarra/Pamplona/Navarra/Spain, Pamplona, Navarre
  - University of Navarra, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: No